CLINICAL TRIAL: NCT02954627
Title: Ultrasound Assessment of the Carotid Intimal Medial Thickness in Obese Subjects Following a Significant Weight Loss
Brief Title: Ultrasound Assessment of the Carotid Intimal Medial Thickness in Obese Subjects; Weight Loss
Acronym: CIMT-LOSEIT-I
Status: Completed | Type: Observational
Sponsor: Henrik Gudbergsen (Other)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Organization: Parker Research Institute (Other)
Other Study IDs: 137.09
Record Dates: First submitted 2016-10-28; First posted 2016-11-03 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis; Obesity
Keywords: Osteoarthritis; Obesity; Liraglutide 3 mg; Liraglutide; Ultrasound
MeSH Terms: conditions — Osteoarthritis; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intensive dietary intervention: Supervised dietary weight loss program lasting 8 weeks
  Interventions: Dietary Supplement: Dietary Supplement: Intensive dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Intensive dietary intervention — Participants receive a hypo-caloric formula diet containing 800 to 1,000 kcal/day. The formula diet consists of ready-to-use meal bars and powders to mix with water to make shakes, soups, or porridge. The weight loss programme consists of an 8-week period with full meal replacement by a standard liquid energy intake protocol. To facilitate compliance with the programme, participants will be scheduled for weekly facility-based group sessions with 6-8 participants led by a dietician. The recommendations for daily nutrient intake will be met.

SUMMARY:
This is a substudy to a randomised trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis (NCT02905864). In the parent trial, patients will be subjected to an 8-week diet intervention phase including a low-calorie diet and dietetic counseling, after which patients will be randomised to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

This substudy aims to investigate any changes in the carotid intima media thickness (CIMT) assessed by ultrasound in relation to an initial 8-week weight loss intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Clinical diagnosis of knee OA (American College of Rheumatology (ACR) criteria) confirmed by radiology but restricted to definite radiographic OA at early to moderate-stages (Kellgren-Lawrence grades 1, 2, or 3)
* Age ≥ 18 years and < 75 years
* Body mass index (BMI) ≥ 27 kg/m2
* Stable body weight during the previous 3 months (< 5 kg self-reported weight change)
* Motivated for weight loss

Exclusion Criteria:

* On-going participation, or participation within the last 3 months, in an organised weight loss programme (or within the last 3 months)
* Current or history of treatment with medications that may cause significant weight gain for at least 3 months before this trial
* Current use or use within three months before this trial of GLP-1 receptor agonist, pramlintide, sibutramine, orlistat, zonisamide, topiramate, or phentermine
* Type 1 diabetes
* Type 2 diabetes treated with glucose-lowering drugs other than metformin
* Alloplasty in target knee joint (see section 6.3)
* End stage disease in target knee joint (Kellgren-Lawrence grade 4)
* Immuno-inflammatory disease
* Chronic wide-spread pain
* Pregnancy or insufficient anti-conception therapy for female fertile patients
* Breast-feeding
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x above upper normal range (UNR)
* Surgery scheduled for the trial duration period, except for minor surgical procedures
* Surgical procedures such as arthroscopy or injections into a knee within 3 months prior to enrolment
* Previous surgical treatment for obesity (excluding liposuction >1 year before trial entry)
* Thyroid stimulating hormone (TSH) outside of the range of 0.4-6.0 mIU/L
* Obesity secondary to endocrinologic or eating disorders or to treatment with medicinal products that may cause weight gain
* Family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Inflammatory bowel disease
* Congestive heart failure, New York Heart Association (NYHA) class III-IV
* Diabetic gastroparesis
* History of or current diagnosis of pancreatitis (acute and/or chronic) or pancreatic cancer
* History of cancer with the exception of in-situ malignancies of the skin or cervix uteri
* History of major depressive disorder, a PHQ-9 (Patient Health Questionnaire-9) score of more than 15, or a history of other severe psychiatric disorders or diagnosis of an eating disorder
* Subjects with a lifetime history of a suicide attempt or history of any suicidal behaviour within the past month before entry into the trial
* Inability to speak Danish fluently
* A mental state impeding compliance with the program
* Use of opioids or similar strong analgesics
* Allergic reactions to the active ingredients of Saxenda, such as hypotension, palpitations, dyspnoea and oedema

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants eligible for parent trial (NCT02905864), i.e. overweight/obese individuals with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in the mean posterior wall common carotid intima-media thickness in mm | Week -8 to 0
  Change will be assessed by grey-scale ultrasound of the posterior wall of the common carotids (one position)
Change in the mean posterior wall common carotid intima-media thickness in mm | Week -8 to 52
  Change will be assessed by grey-scale ultrasound of the posterior wall of the common carotids (one position)

SECONDARY OUTCOMES:
Change in the maximum posterior wall common carotid intima-media thickness in mm | Week -8 to 0
  Change will be assessed by grey-scale ultrasound of the posterior wall of the common carotids (one position)
Change in the maximum posterior wall common carotid intima-media thickness in mm | Week -8 to 52
  Change will be assessed by grey-scale ultrasound of the posterior wall of the common carotids (one position)

CONTACTS AND LOCATIONS:
Locations (1):
- Osteoarthritis Clinic, Frederiksberg, Capital Region, Denmark